CLINICAL TRIAL: NCT00047736
Title: A Phase III, Randomized, Double Blind, Multicenter Trial of Tarceva (Erlotinib) Plus Chemotherapy (Carboplatin and Paclitaxel) Versus Chemotherapy Alone in Patients With Advanced (Stage IIIb or IV) Non-Small Cell Lung Cancer Who Have Not Received Prior Chemotherapy
Brief Title: A Study With Tarceva and Chemotherapy vs. Chemotherapy Alone in Patients With Advanced Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: OSI2298g; NCT00029016 (obsolete NCT alias)
Record Dates: First submitted 2002-10-16; First posted 2002-10-17 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Tarceva (erlotinib HCl)

SUMMARY:
The purpose of this study is to determine if Tarceva plus standard chemotherapy is more effective than standard chemotherapy alone in the treatment of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >=18 years
* Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic Stage IIIB or Stage IV Non-Small Cell Lung Cancer (NSCLC)
* A cytologic diagnosis is acceptable (i.e., FNA or pleural fluid cytology)
* Measurable or non-measurable disease
* ECOG performance status of 0 or 1
* Life expectancy of >=3 months
* >= 3 weeks since any prior surgery or radiotherapy (>=2 weeks for patients who receive <=30 Gy of radiotherapy involving <25% of the marrow reserve)
* Use of an effective means of contraception (women of childbearing potential)
* Able to comply with study and follow-up procedures

Exclusion Criteria:

* Evidence of small cell, carcinoid, or mixed small cell/non-small cell histology
* Malignancies within 3 years except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
* Symptomatic or untreated brain metastases
* Prior systemic chemotherapy for NSCLC
* Prior exposure to agents directed at the HER axis (e.g., ZD1839 [Iressa], C225 [Cetuximab], Trastuzumab [Herceptin])
* Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or serious cardiac arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible)
* History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption
* Pregnancy or lactation

Any of the following abnormal baseline hematologic values:

* Granulocytes count <=1500/uL
* Platelet count <100,000/uL

Any of the following abnormal baseline liver function tests:

* Serum bilirubin >1.5× upper limit of normal (ULN)
* Serum ALT and AST >=2.5× ULN (>5× ULN if due to liver metastases)
* Alkaline phosphatase >=2.5× ULN

Other baseline laboratory values:

* Serum creatinine >1.5× ULN or creatinine clearance <60 mL/min
* Uncontrolled hypercalcemia (>11.5 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Multinational Sites, Denver, Colorado
  - Trial Information Center, Denver, Colorado

REFERENCES:
- [Result] Hirsch FR, Varella-Garcia M, Dziadziuszko R, Xiao Y, Gajapathy S, Skokan M, Lin M, O'Neill V, Bunn PA Jr. Fluorescence in situ hybridization subgroup analysis of TRIBUTE, a phase III trial of erlotinib plus carboplatin and paclitaxel in non-small cell lung cancer. Clin Cancer Res. 2008 Oct 1;14(19):6317-23. doi: 10.1158/1078-0432.CCR-08-0539. PMID 18829515